CLINICAL TRIAL: NCT05929755
Title: Effect of Depo-Medrol Application on the Psoas Muscle After Transpsoas LLIF on Post-operative Hip Flexor Weakness, Thigh Pain and Numbness
Brief Title: Depo-Medrol on Psoas After LLIF
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hardeep Singh (Other)
Collaborators: Society for Minimally Invasive Spine Surgery (Other)
Responsible Party: Sponsor-Investigator, Hardeep Singh, Assistant Professor of Orthopedic Surgery, UConn Health
Organization: UConn Health (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 23-090-2
Record Dates: First submitted 2023-05-26; First posted 2023-07-03 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Muscle Weakness; Pain, Postoperative; Paresthesia; Pain, Muscle
Keywords: lateral lumbar interbody fusion; LLIF; Depo-Medrol; corticosteroid; lumbar spine; psoas muscle; postoperative hip flexor weakness; postoperative thigh pain; postoperative thigh numbness
MeSH Terms: conditions — Muscle Weakness; Pain, Postoperative; Paresthesia; Myalgia | interventions — Methylprednisolone Acetate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (standard care) (Placebo Comparator): 1 cc gel foam powder mixed with thrombin
  Interventions: Drug: Gel-Flow NT
- Test group (standard care + study intervention) (Experimental): 1 cc of gel foam powder mixed with thrombin and 80mg Depo-Medrol
  Interventions: Drug: Depo-Medrol; Drug: Gel-Flow NT

INTERVENTIONS:
Drug: Depo-Medrol — steroid
  Arms: Test group (standard care + study intervention)
Drug: Gel-Flow NT — hemostatic agent

SUMMARY:
The goal of this study is to determine the effects of a corticosteroid administered to the psoas muscle following a transpsoas lateral lumbar interbody fusion (LLIF) on postoperative hip flexor weakness and thigh pain and numbness.

DETAILED DESCRIPTION:
Primary Objective and Outcome Measure:

* Quantify the difference in thigh pain measured on the visual analog pain scale (VAS) between those receiving a depo-medrol injection and those who did not over 3 postoperative time periods: 2-3, 6, and 12 weeks following surgery.

Secondary Objectives and Outcome Measures:

* Quantify the difference in rates and severity of postoperative hip flexor weakness, and numbness both with and with out application of depo-medrol to the psoas between those that did and did not receive a depo-medrol injection.
* Quantity patient reported outcomes measures (PROMs) (EQ5D, ODI, and sciatica Bothersome index between those that did and did not receive a depo-medrol injection. Specifically:

  * EQ5D: Eur-Quality of Life 5 dimension questionnaire
  * ODI: Oswestry Disability Index
* Determine effect of depo-medrol application on fusion rates and how it differs between those that did and did not receive a depo-medrol injection.

Ancillary Objectives and Outcome Measures:

* To determine the effect of clinically relevant covariates including sociodemographic and comorbidities on the course of postoperative pain and associated outcome measures and whether the effect of these covariates moderate the effect of postoperative pain.

Groups:

* Control group (standard care) - 1cc gel foam powder mixed with thrombin
* Steroid group (standard care + study intervention) - 1cc gel foam powder mixed with thrombin and 80mg depomedrol

ELIGIBILITY:
Inclusion Criteria:

* Patients from the practices of Drs. Singh, Mallozzi, Moss
* Transpsoas (PTP or LTP) lateral lumbar interbody fusion (LLIF) 1-3 disc levels with posterior instrumentation (Open or MIS) with or without laminectomy, must include L3-4 and/or L4-5
* Patients who agree to be a part of the study
* Patients with lumbar disc degeneration
* Patients between ages of 18 and 75

Exclusion Criteria:

* Scoliosis >10°
* Spondylolisthesis >Grade 1
* Flatback deformity
* Patients with insulin dependent diabetes
* Patients with >3 levels of fusion
* Alternative interbodies
* Chronic oral steroid users
* Patients with allergy/intolerance to depo-medrol or other steroids
* Patients requiring bilateral transpsoas approaches
* Patients with ipsilateral symptomatic hip pathology
* Revision fusion procedures
* Cases involving trauma, tumor, or infection
* Patient's not capable of providing consent themselves
* Non-fluent English speakers (for consenting reasons)
* Patients who are lost to follow-up before the two year follow up period

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-05-12 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Quantify the difference in thigh pain measured on the visual analog pain scale (VAS) between those receiving a depo-medrol injection and those who did not over 3 postoperative time periods: 2-3, 6, and 12 weeks following surgery. | 2-3 weeks following surgery
  Visual Analog Scale (VAS) - Anterior Thigh Pain
  How would you evaluate the pain you are feeling today at the front of your thigh on a scale from "no pain" to "worst pain imaginable"?
Quantify the difference in thigh pain measured on the visual analog pain scale (VAS) between those receiving a depo-medrol injection and those who did not over 3 postoperative time periods: 2-3, 6, and 12 weeks following surgery. | 6 weeks following surgery
  Visual Analog Scale (VAS) - Anterior Thigh Pain
  How would you evaluate the pain you are feeling today at the front of your thigh on a scale from "no pain" to "worst pain imaginable"?
Quantify the difference in thigh pain measured on the visual analog pain scale (VAS) between those receiving a depo-medrol injection and those who did not over 3 postoperative time periods: 2-3, 6, and 12 weeks following surgery. | 12 weeks following surgery
  Visual Analog Scale (VAS) - Anterior Thigh Pain
  How would you evaluate the pain you are feeling today at the front of your thigh on a scale from "no pain" to "worst pain imaginable"?

SECONDARY OUTCOMES:
Quantify the difference in rates of postoperative thigh numbness both with and with out application of depo-medrol to the psoas between those that did and did not receive a depo-medrol injection. | 6 months, 1 year, 2 years
  Thigh numbness - binary: yes/no
Quantify the difference in severity of postoperative hip flexor weakness both with and with out application of depo-medrol to the psoas between those that did and did not receive a depo-medrol injection. | 6 months, 1 year, 2 years
  Hip flexion strength measured via graded exam: the Medical Research Council Manual Muscle Testing scale. This method involves testing key muscles from the lower extremities against the examiner's resistance and grading the patient's strength on a 0 to 5 scale accordingly:
  0 No muscle activation
  1. Trace muscle activation, such as a twitch, without achieving full range of motion
  2. Muscle activation with gravity eliminated, achieving full range of motion
  3. Muscle activation against gravity, full range of motion
  4. Muscle activation against some resistance, full range of motion
  5. Muscle activation against examiner's full resistance, full range of motion
Quantity patient reported outcomes measures (PROMs) between those that did and did not receive a depo-medrol injection: Euro-Quality of Life 5 dimension questionnaire (EQ5D) | 2-3 weeks, 6 weeks, 12 weeks, 6 months, 1 year, and 2 years
  The Euro-Quality of Life 5 Dimension 5 Level (EQ-5D-5L) is a self-report survey that measures quality of life across 5 domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is scored on a 5-level severity ranking that ranges from "no problems" through "extreme problems."
Quantity patient reported outcomes measures (PROMs) between those that did and did not receive a depo-medrol injection: Oswestry Disability Index (ODI) | 2-3 weeks, 6 weeks, 12 weeks, 6 months, 1 year, and 2 years
  The Oswestry Disability Index (ODI) is an outcome measure that was designed to assess function in activities of daily living for those with acute or chronic back pain. The ODI consists of 10 patient-completed questions in which the response options are presented as 6-point Likert scales. Scores range from 0% (no disability) to 100% (most severe disability).
Quantity patient reported outcomes measures (PROMs) between those that did and did not receive a depo-medrol injection: Sciatica Bothersomeness Index | 2-3 weeks, 6 weeks, 12 weeks, 6 months, 1 year, and 2 years
  Sciatica Bothersomeness index includes self-reported ratings of symptom intensity of:
  * Leg pain
  * Numbness or tingling in the leg, foot or groin
  * Weakness in the leg/foot
  * Back or leg pain while sitting
  Each symptom item is rated on a scale from 0 to 6, with 0 being not bothersome, 3 somewhat bothersome and 6 extremely bothersome.
Determine effect of depo-medrol application on fusion rates and how it differs between those that did and did not receive a depo-medrol injection. | 1 year and 2 years
  Fusion rate - Assessed with Flexion, Extension X-ray (screw loosening/fracture, instability)
  CT Scan if patient has a symptomatic (pain) pseudoarthrosis (lack of fusion)

CONTACTS AND LOCATIONS:
Overall Officials: Hardeep Singh, M.D., Principal Investigator — UConn Health
Locations (1):
- UConn Health, Farmington, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No